CLINICAL TRIAL: NCT03278392
Title: Prenatal Emotion-Diet Interactions and the Metabolic Response
Brief Title: Maternal Emotions and Diet in Pregnancy
Acronym: PEDIMet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, San Francisco (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Karen Lindsay, Principal Investigator, University of California, Irvine
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UCI 2017-3803
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Pregnancy Related; Stress, Psychological; Glucose Intolerance During Pregnancy
Keywords: pregnancy; metabolism; stress; emotional state; diet; glycemic response
MeSH Terms: conditions — Stress, Psychological | interventions — Psychological Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial challenge task (Experimental): Participants will be assigned to complete the Trier Social Stress Test (TSST) immediately after consuming a standardized breakfast drink
  Interventions: Behavioral: Trier Social Stress Test
- Placebo challenge task (Sham Comparator): Participants will be assigned to complete the placebo non-stress task immediately after consuming a standardized breakfast drink
  Interventions: Behavioral: Placebo Non-stress task

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Task instructions provided to subject (5mins), subject prepares speech on their strengths and weaknesses (5 mins), subject delivers speech before a stern evaluative committee while being video-taped (5 mins), subject completes a mental arithmetic challenge task before the evaluative committee with critiques if errors are made (5mins).
  Arms: Psychosocial challenge task
Behavioral: Placebo Non-stress task — Subject engages in a friendly conversation about a neutral or happy topic (e.g. recent holiday, favorite past-times) for 15 minutes with a familiar research staff member.
  Arms: Placebo challenge task

SUMMARY:
This study seeks to understand how a mother's emotional state in pregnancy influences her biological response to food intake.

DETAILED DESCRIPTION:
The purpose of this research study is to understand how a mother's emotional state in pregnancy influences her biological response to food intake. Natural variation in emotional and mental state is frequently experienced in daily life, including during pregnancy. While the investigators understand that a healthy diet is important in pregnancy for maintaining blood sugar levels and other metabolic factors within normal ranges for optimal development of the baby, less consideration is given to the health effects of a mother's mental state during pregnancy. It may even be possible that, regardless of what a woman eats or drinks, the way her body responds to food may differ according to her emotional or mental state.

This research is particularly interested in understanding how the combination of maternal emotional state and diet influence metabolism in pregnancy. Thus, the aim of this study is to test whether and how an individual's emotional response to a mental challenge of varying complexity during pregnancy modifies the body's metabolic response to a standard breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Hispanic ethnicity
* English and/or Spanish speaking
* Multiparous
* 28-30 week's gestation
* Pre-pregnancy BMI 25.0-34.9 kg/m2
* Singleton, intrauterine pregnancy
* Non-smoker
* Non-diabetic and negative result on routine prenatal glucose challenge test (GCT)

Exclusion Criteria:

* BMI <25.0 or ≥35.0 kg/m2
* >30 week's gestation
* multiple pregnancy
* nulliparous
* present/prior obstetric risk conditions (hypertension, preeclampsia, infections, placental abnormalities)
* current smoker
* current psychiatric disorders or undergoing treatment/taking psychiatric medications
* Use of systemic/frequent corticosteroids or thyroid meds
* Diabetic or presence of other metabolic or neuroendocrine disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Difference in the glycemic response to the standardized meal +/- psychosocial challenge task | 2 hours
  Glycemic response (area-under-the-curve of glucose) to the standardized breakfast drink following exposure to either the psychosocial challenge (TSST) or non-challenge (placebo-TSST) task.

SECONDARY OUTCOMES:
Difference in the triglyceride response to the standardized meal +/- psychosocial challenge task | 2 hours
  Area under the curve of blood triglycerides to the standardized breakfast drink following exposure to either the psychosocial challenge (TSST) or non-challenge (placebo-TSST) task.
Physiological stress response to the psychosocial challenge task | 2 hours
  Area under the curve of salivary cortisol following exposure to the psychosocial challenge task

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Lindsay, Principal Investigator — UC Irvine
Locations (1):
- UCI Medical Center, University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindsay KL, Buss C, Wadhwa PD, Entringer S. The Interplay between Maternal Nutrition and Stress during Pregnancy: Issues and Considerations. Ann Nutr Metab. 2017;70(3):191-200. doi: 10.1159/000457136. Epub 2017 Mar 17. PMID 28301838